CLINICAL TRIAL: NCT03783793
Title: Effects of a Mindfulness Meditation App on Subjective Well-Being: Active Randomized Controlled Trial and Experience Sampling Study
Brief Title: Effects of a Mindfulness Meditation App on Subjective Well-Being in Undergraduate University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario centre for excellence vip program (Unknown)
Responsible Party: Principal Investigator, Norman Farb, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32099
Record Dates: First submitted 2018-12-14; First posted 2018-12-21 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Stress, Psychological
Keywords: mindfulness; attention; mobile health; interoception; mood
MeSH Terms: conditions — Stress, Psychological | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training App (Experimental)
  Interventions: Behavioral: Mindfulness Training App
- Cognitive Training With 2048 (Active Comparator)
  Interventions: Behavioral: Cognitive Training With 2048

INTERVENTIONS:
Behavioral: Mindfulness Training App — Mindfulness training in the study was performed using a new app called Wildflowers. With this app participants were able to choose and complete a variety of guided meditations over the 3 week training period. Wildflowers includes guided meditations such as breathing, body scans, and open monitoring practices and also provides didactic content in the form of lessons and information about the benefits of mindfulness training.
  Arms: Mindfulness Training App
Behavioral: Cognitive Training With 2048 — The training app for the control condition was based on an open source code for a popular cognitive training app called 2048 that is marketed as a fun and relaxing puzzle game. Within 2048, participants slide numbered tiles around a grid, matching tiles of the same value. Instead of tiles disappearing, as in Candy Crush or other similar grid-sliding games, matching 2 numbered tiles in 2048 combines them into 1 new tile displaying the sum of the previous 2 numbers. For example, two 2-tiles linked side-by-side become a 4-tile, whereas 2 matched 4-tiles become an 8-tile, and so on. The goal is to match tiles until the sum of 2048 is reached on a single tile. There is no time limit.
  Arms: Cognitive Training With 2048

SUMMARY:
Mindfulness training includes a variety of contemplative practices aimed at promoting intentional awareness of experience, coupled with attitudes of non-judgment and curiosity. Following the success of 8-week, manualized group interventions, mindfulness training has been implemented in a variety of modalities, including smartphone apps that seek to replicate the success of group interventions. However, although smartphone apps are scalable and accessible to a wider swath of population, their benefits remain largely untested. This study aimed to investigate a newly developed mindfulness training app called Wildflowers, which was co-developed with the laboratory for use in mindfulness research. It was hypothesized that 3 weeks of mindfulness training through this app would improve subjective well-being, attentional control, and interoceptive integration, albeit with weaker effects than those published in the 8 week, manualized group intervention literature.

DETAILED DESCRIPTION:
Background: Mindfulness training includes a variety of contemplative practices aimed at promoting intentional awareness of experience, coupled with attitudes of non-judgment and curiosity. Following the success of 8-week, manualized group interventions, mindfulness training has been implemented in a variety of modalities, including smartphone apps that seek to replicate the success of group interventions. However, although smartphone apps are scalable and accessible to a wider swath of population, their benefits remain largely untested. This study aimed to investigate a newly developed mindfulness training app called Wildflowers, which was co-developed with the laboratory for use in mindfulness research. It was hypothesized that 3 weeks of mindfulness training through this app would improve subjective well-being, attentional control, and interoceptive integration, albeit with weaker effects than those published in the 8 week, manualized group intervention literature.

Methods: Undergraduate students completed 3 weeks of mindfulness training with Wildflowers or 3 weeks of cognitive training with a game called 2048. State training effects were assessed through pre- and postsession ratings of current mood, stress level, and heart rate. Trait training effects were assessed through pre- and postintervention questionnaires canvassing subjective well-being and behavioral task measures of attentional control and interoceptive integration. State and trait training data were analyzed in a multilevel model using emergent latent factors (acceptance, awareness, and openness) to summarize the trait questionnaire battery.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision and hearing
* Be fluent in english
* Own an iPhone, iPad, or iPod with access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Change on the Perceived Stress Scale | 0 weeks and 3 weeks
  A 4-item self-report scale that measures the global perception of stress. The scale asks participants about their feelings and thoughts during the last month, and participants indicate on a 5-point Likert scale how often they thought or felt a certain way, with 0 being never and 4 being very often. A higher score on this measure represents higher levels of self-reported stress (worse outcome) with a minimum possible score of 0 and a maximum of 16.
Change on the Big Five Inventory | 0 weeks and 3 weeks
  A 44-item self-report scale that measures the 5 dimensions of personality: extraversion, agreeableness, conscientiousness, neuroticism, and openness. On this scale, participants are asked if different characteristics apply to them. For each characteristic queried participants respond on a 5-point Likert scale, with 1 being disagree strongly and 5 being agree strongly. This scale yields 5 scores, one for each of the subscales: extraversion (min-max range: 8-40), agreeableness (min-max range: 9-45), conscientiousness (min-max range: 9-45), neuroticism (min-max range: 8-40), and openness (min-max range: 10-50). Higher values on each of the subscales represent higher levels of that particular personality trait.
Change on the Psychological Well-Being Scale | 0 weeks and 3 weeks
  An 84-item self-report questionnaire that measures psychological well-being. Respondents rate statements on a 6-point likert scale, with 1 being strong disagreement and 6 being strong agreement. This measure yields 6 scores, one for each subscale: autonomy, self-acceptance, positive relations with others, environmental mastery, purpose in life, and personal growth. Each of these subscales have a possible minimum score of 14 and a maximum score of 84 with higher values representing a better outcome.
Change on the Acceptance and Action Questionnaire-II | 0 weeks and 3 weeks
  A 7-item self-report scale that measures psychological inflexibility and experiential avoidance. Respondents rate a list of statements on a 7-point likert scale, with 1 being never true and 7 being always true. This measure yields one score with a possible minimum of 7 and a maximum of 49. Higher values represent greater levels of psychological inflexibility (worse outcome).
Change on the Philadelphia Mindfulness Scale | 0 weeks and 3 weeks
  A 20-item self-report scale that measures 2 components of mindfulness: awareness and acceptance. Respondents rate a series of statements on a 5-point likert scale, with 1 being never and 5 being very often. This scale yields two scores, one for each subscale: awareness and acceptance. On the awareness scale the minimum possible score is 10 and the maximum is 50. Higher values on this subscale represent higher levels of awareness (better outcome). For the acceptance subscale, the minimum possible score is 10 and the maximum is 50, with higher values representing higher levels of acceptance (better outcome).
Change on the Multidimensional Assessment of Interoceptive Awareness | 0 weeks and 3 weeks
  A 32-item self-report scale that measures the multidimensional construct of interoceptive body awareness. Respondents rate a list of statements on a 6-point likert scale, with 0 being never and 5 being always. This measure yields 8 scores, one for each of the subscales: noticing (min-max range: 0-20), not distracting (min-max range: 0-15), not worrying (min-max range: 0-15), attention regulation (min-max range: 0-35), emotional awareness (min-max range: 0-25), self-regulation (min-max range: 0-20), body listening (min-max range: 0-15), and trusting (min-max range: 0-15). On each of these subscales, higher values represent higher levels of interoceptive body awareness (better outcome).
Change on the Spiritual Experience Index-Revised | 0 weeks and 3 weeks
  A 23-item self-report scale that measures a person's faith and spiritual journey. Respondents rate a list of statements on a 6-point likert scale, with 1 being strongly disagree and 6 being strongly agree. This measure yields two scores, one for each subscale: spiritual support (min-max range: 13-78) and spiritual openness (min-max range: 10-60). On the spiritual support subscale, higher values represent higher levels of spiritual support (better outcome). On the spiritual openness subscale, higher values represent higher levels of spiritual openness (better outcome).
Change on the Meaning in Life Questionnaire | 0 weeks and 3 weeks
  A 10-item self-report scale that measures 2 dimensions of the meaning in life and as such includes 2 subscales: presence of meaning and search for meaning. Respondents rate statements on a 7-point Likert scale, with 1 being absolutely untrue and 7 being absolutely true. On the presence of meaning subscale the minimum possible score is 5 and the maximum is 35, with higher values representing the degree that participants feel they have meaning in their lives (better outcome). On the search for meaning subscale the minimum possible score is 5 and the maximum is 35, with higher values representing the extent that individuals are searching for meaning in their lives (better outcome).
Change on the Mood Board Circumplex | 0 weeks and 3 weeks
  The mood board is a visual representation of negative and positive emotions on a spectrum, ranging from intense emotions to mild emotions. This mood board provides a maximum of 32 emotions that a participant can select by clicking on that emotion. This measure yields 4 scores one for each subscale. Each subscale has a minimum possible score of 0 and maximum of 8. Higher values on the intense negative emotions subscale represent greater levels of intense negative emotions (worse outcome). Higher values on the intense positive emotions subscale represents greater levels of intense positive emotions (better outcome). Higher values on the mild negative emotions subscale represents greater levels of mild negative emotions (worse outcome). Lastly, higher values on the mild positive emotions subscale represents greater levels of mild positive emotions (better outcome).
Change on the Centre for Research on Safe Driving-Attention Network Test | 0 weeks and 3 weeks
  This is a 10-min version of the Attention Network Test that measures 3 different functions of attention:
  alerting, orienting, and conflict monitoring.
Change on the Respiration Integration Task | 0 weeks and 3 weeks
  This is a newly developed behavioral task created in our laboratory to assess interoceptive attention.
Change in Mood | 0 minutes and approximately 10 minutes, every day for 3 weeks.
  Mood was measured via self-report on the smartphone app. This measurement was taken before and after each use of the smartphone app in their assigned condition.
Change in Stress | 0 minutes and approximately 10 minutes, every day for 3 weeks.
  Stress was measured using a visual analogue scale on a smartphone app where participants would rate their level of stress by sliding a bar along the scale. They would slide the bar to the green side of the scale if experiencing low levels of stress and to the red side of the scale if experiencing high levels of stress. This is a continuous scale with a minimum possible score of 0 and a maximum score of 1, with higher values representing greater levels of stress (worse outcome). This measurement was taken before and after each use of the smartphone app in their assigned condition.
Change in Heart Rate | 0 minutes and approximately 10 minutes, every day for 3 weeks.
  Heart rate was measured using the camera on the smartphone app using a well established algorithm. This measurement was taken before and after each use of the smartphone app in their assigned condition.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walsh KM, Saab BJ, Farb NA. Effects of a Mindfulness Meditation App on Subjective Well-Being: Active Randomized Controlled Trial and Experience Sampling Study. JMIR Ment Health. 2019 Jan 8;6(1):e10844. doi: 10.2196/10844. PMID 30622094